CLINICAL TRIAL: NCT05485155
Title: An Open-Label Study of Zemaira (Alpha 1-Trypsin Inhibitor) in Subjects With Eosinophilic Esophagitis
Brief Title: Zemaira Eosinophilic Esophagitis Pilot Study
Acronym: ZEEPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: CSL Behring (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0625
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Active Drug (Experimental): Zemaira alpha-proteinase inhibitor
  Interventions: Drug: Alpha-proteinase inhibitor

INTERVENTIONS:
Drug: Alpha-proteinase inhibitor — Intravenous infusion at 120 mg/kg body weight dose/week for 4 weeks for a total of 4 infusions.
  Other Names: Zemaira

SUMMARY:
This is a prospective, open-label drug study that will examine the effects of Zemaira (alpha-1 trypsin inhibitor) in patients with Eosinophilic Esophagitis.

DETAILED DESCRIPTION:
This is a phase II, open-label trial of Zemaira in participants diagnosed with eosinophilic esophagitis. Potential participants will be screened during a 12-week screening period. Participants will be enrolled based on the presence of active disease and their ability to meet the study inclusion and exclusion criteria. Qualifying participants will receive weekly intravenous infusions of 120 mg/kg body weight dose/week for 4 weeks (for a total of 4 infusions). During the treatment period, participants will be monitored for adverse events/reactions and will complete patient reported outcome metrics to track their symptoms and general wellbeing. Final assessments will be performed 24 hours after the last dose of the study drug. All participants will be followed for an additional 12 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or legally authorized representative must be able to understand and provide informed consent prior to study procedures being performed.
2. Willing and able to comply with study visits and activities
3. Age ≥ 18 to ≤ 70 years at study enrollment
4. Histologically active eosinophilic esophagitis (EoE) at time of screening or within 12 weeks prior to enrollment, with a peak count of ≥ 15 eosinophils (eos)/high powered field (hpf) in any region of the esophagus, with no other known cause for esophageal eosinophilia; involvement of eosinophilic inflammation in other gastrointestinal segments will be allowed but not required or sufficient.
5. History of approximately 8 week standard of care (SOC) treatment (e.g., proton pump inhibitors (PPI's), topical corticosteroids) that did not adequately control or treat the EoE or documentation that such treatment was not tolerated. Participant may re-screen if this is not met.
6. Stable medical management of EoE (and other eosinophilic disorders, if applicable) including stable dosage of medications in the 8 weeks prior to study enrollment, if applicable. Participants may be on baseline anti-EoE therapy (such as elimination diet, elemental diet, proton pump inhibitors (PPI), topical or systemic glucocorticoids (≤10 milligrams (mg) daily), immunosuppressive agents, cromolyn, and H1 and H2 anti-histamines) as long as there is agreement not to change their dosage.
7. Willing to maintain current dietary regimen throughout the course of the study. Diet must have been stable for 8 weeks prior to baseline endoscopy.

Exclusion Criteria:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
2. Current active H. pylori infection. A history of H. pylori infection needs to have medical documentation of one of the three acceptable eradication tests: antigen, breath or histology. Participants with current active H. pylori infections can be re-screened for study participation in the future if they are treated and have medical documentation of one of the three acceptable eradication tests: antigen, breath or histology.
3. Another disorder that causes esophageal eosinophilia (e.g., hypereosinophilic syndrome*, Churg Strauss vasculitis, eosinophilic granuloma or a parasitic infection).

   *Hypereosinophilic syndrome defined by multiple organ involvement (with the exception of atopic disease or eosinophilic gastrointestinal disorder (EGID)) and persistent blood absolute eosinophil count ≥1500/microliter.
4. Systemic gastrointestinal disorders such as Crohn's disease, inflammatory bowel disease, or Celiac disease not including chronic gastritis, chronic duodenitis, mucosal eosinophilia or other EGID's.
5. Diagnosed with Chronic Obstructive Pulmonary Disease (COPD).
6. Known immunoglobulin A (IgA) deficiency (i.e., IgA level < 8 mg/dL at screening).
7. Current coronavirus disease of 2019 (COVID-19) infection (i.e., detection of the presence of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) before the screening endoscopy using testing done at the clinical site).
8. Hematological disorders that prevent the blood from clotting (e.g., hemophilia, Von Willebrand disease, clotting factor deficiencies).
9. Currently on anti-coagulation medications (except aspirin/Non-steroidal anti-inflammatory drugs).
10. Known history of hypersensitivity following infusions of human blood or blood components (e.g., human immunoglobulins or human albumin).
11. Known history of hypersensitivity or anaphylaxis to Zemaira or other A1AT products.
12. Uncontrolled, or poorly controlled, comorbid conditions including, but not limited to, cardiovascular diseases, hypertension and diabetes as defined by the following criteria:

    * A myocardial infarction within the last 6 months.
    * Blood pressure > 179/99 mmHg
    * Diabetics with a hemoglobin A1C (HbA1C) > 7% and that are deemed to have uncontrolled diabetes as defined by the physician
13. History of cancer: Individuals who have had basal cell carcinoma, localized squamous cell carcinoma of the skin, or in situ carcinoma of the cervix are eligible provided that the participant is in remission and curative therapy was completed at least 12 months prior to the date informed consent was obtained. Individuals who have had other malignancies are eligible provided that the individual is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained.
14. Current or recent use of any investigational drug (within 3 months or 5 half-lives, whichever is longer, prior to screening).
15. Currently participating or planning to participate in another clinical study involving an investigational drug during the course of this study.
16. Presence of steroid-responsive diseases (e.g., asthma) with a recent (within the last 6 months) history of disease exacerbations requiring steroid treatment.
17. Current use of systemic steroids with daily dose > 10 mg for any reason or steroid burst for > 3 days within 1 month of screening.
18. Current pregnancy or breastfeeding.
19. Any esophageal stricture unable to be passed with a standard, diagnostic upper endoscope.
20. Esophageal varices or interventional treatment for esophageal varices that, in the opinion of the investigator, would put the participant at undue risk for significant complications from an endoscopy procedure.
21. History of alcohol or drug abuse within 6 months prior to screening.
22. Participant or his/her immediate family is a member of the investigational team.
23. Presence of clinically significant laboratory abnormalities at the screening that meets one or more of the following criteria:

    1. Serum alanine aminotransferase (ALT) ≥ 3 times upper limit of normal (ULN)
    2. Serum total bilirubin ≥2 times ULN
    3. Absolute neutrophil count (ANC) ≤ 1000 cells/mm3
    4. Hemoglobin (Hgb) ≤ 10.0 g/dL
    5. Platelet count ≤ 100,000/mm3
    6. Glomerular Filtration Rate (GFR) ≤ 44 mL/min/1.73 m2
24. Planned or anticipated major surgical procedure during the study.
25. Known or suspected immunodeficiency disorder, including human immunodeficiency disorder (HIV) or a history of invasive opportunistic infections (e.g., tuberculosis, non-tuberculous mycobacterial infections, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis, or an infectious etiology of esophagitis (e.g. cytomegalovirus or Candida) despite infection resolution or otherwise recurrent infections of abnormal frequency or prolonged infections suggesting an immune-compromised status as judged by the investigator.
26. Planned or anticipated use of any prohibited medications and procedures during the study.
27. Currently on Zemaira for other indications.
28. Initiation, discontinuation or change in the dosage regimen of the following medications within 8 weeks prior to the baseline endoscopy:

    Proton pump inhibitors Leukotriene inhibitors Nasal and/or inhaled corticosteroids Participants on a stable dose of these medications for at least 8 weeks prior to the baseline endoscopy may be included in the study. PPI and leukotriene inhibitor dosing must not change during the study, but nasal and/or inhaled corticosteroids can be increased if there is a deterioration in the condition for which the medications are prescribed.
29. Presence of the following esophageal disorders: achalasia cardia, Barrett's esophagus or precancerous lesions noted on the endoscopy.
30. Women of childbearing potential, or male participants with female partners of childbearing potential, who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment, during the study, and for at least 12 weeks after the last dose. Highly effective contraceptive measures include:

    1. Stable use of combined (estrogen and progestogen containing) hormonal contraception (oral, intravaginal, transdermal) or progestogen-only hormonal contraception (oral, injectable, implantable) for one month prior to screening
    2. Intrauterine device; intrauterine hormone-releasing system
    3. Bilateral tubal ligation
    4. Vasectomized partner
    5. And/or sexual abstinence
31. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in esophageal alpha1 anti-trypsin (A1AT) concentration | 4 weeks
  Absolute change from baseline A1AT esophageal concentration in participants receiving Zemaira to 24 hours after the last infusion at 4 weeks
Adverse events | 20 weeks
  The number of Adverse Events (AE), including Serious Adverse Events (SAE), related to the study drug.

SECONDARY OUTCOMES:
Change in serine protease activity | 4 weeks
  Absolute change from baseline serine protease activity in participants receiving Zemaira to the end of treatment visit at 4 weeks as determined by protease activity testing.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rothenberg, Principal Investigator — Cincinnati Children's Hospital Medical Center
Locations (2):
- United States (2):
  - The National Institutes of Health, Bethesda, Maryland
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No